CLINICAL TRIAL: NCT05109221
Title: Validity of Ultrasonography in Predicting Difficult Laryngoscopy and Confirming Endotracheal Intubation in Obese Emergency Surgical Patients
Brief Title: Ultrasonography in Predicting Difficult Intubation in Obese Emergency Surgical Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hemmat Amer Mohamed, Minia_ Eygpt, Minia University
Other Study IDs: 99_2021
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Preoperative Ultrasound Assessment of the Upper Airway Can Predict Difficult Laryngscopy in Obese at Emergency Operations
Keywords: ultrasound _difficult intubation _obese _emergency operations
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: ultrasound — using of ultrasound in prediction of difficult intubation in obese surgical patients

SUMMARY:
Validity of ultrasonography in predicting difficult laryngoscopy and confirming endotracheal intubation in obese emergency surgical patients

DETAILED DESCRIPTION:
The aim of the study is to determine whether preoperative ultrasound assessment of of the upper airway can predict difficult laryngscopy in emergency surgical obese patients , by analysis correlations between ultrasound measurements of anterior cervical soft in the upper airway, and the Cormack-Lehane grade. And evaluate its role in confirming the endotracheal placement The secondary objective was to determine whether clinical screening tests are independent predictors of difficult airway.

ELIGIBILITY:
Inclusion Criteria:

* Adult obese patients (BMI>35) of both sex aged from 18 to 60 years undergoing urgent surgeries under general anasthesia with tracheal intubation.

Exclusion Criteria:

* . Patients with removable upper dentures, upper airway pathology, cervical spine fractures, full stomach, maxillofacial trauma or unstable patients and pregnant women will be excluded from the study

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: obese emergency surgical patients
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
prediction of difficult intubation in obese emergency surgical patients by ultrasound | 30minutes
  determine whether preoperative ultrasound assessment of of the upper airway can predict difficult laryngscopy in emergency surgical obese patients , by analysis correlations between ultrasound measurements of anterior cervical soft in the upper airway, and the Cormack-Lehane grade. And evaluate its role in confirming the endotracheal placement

CONTACTS AND LOCATIONS:
Locations (1):
- Hemmat amer mohamed, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

DOCUMENTS (2):
  • Study Protocol (2021-08-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT05109221/Prot_000.pdf
  • Informed Consent Form (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/21/NCT05109221/ICF_001.pdf